CLINICAL TRIAL: NCT05587088
Title: Evaluation of the Safety and Efficacy of Esperanza Extract (Petiveria Alliacea) in Patients With Metastatic Gastrointestinal Tumors and Acute Leukemia
Brief Title: Evaluation of the Safety and Efficacy of Esperanza Extract (PA001)
Acronym: PA001
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario San Ignacio (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PA001
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Neoplasm, Stomach; Gastric Neoplasms Malignant; Pancreatic Neoplasms; Colorectal Neoplasms; Acute Leukemia; Acute Leukemia in Relapse; Acute Leukemia Lymphoid; Acute Myeloid Leukemia; Acute Myeloid Leukemia, in Relapse
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This is a phase Ib/II clinical study that has two phases. In phase Ib, the safety evaluation of the extract of Petiveria alliacea (Esperanza) will be carried out in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach and biliary tract) and patients with newly diagnosed and relapsed acute leukemia. In phase IIb, the safety will continue to be evaluated and the efficacy of the Esperanza extract will be explored in combination with chemotherapy in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach and biliary tract) and patients with newly diagnosed acute leukemias and relapses
Who Masked: Participant, Care Provider, Investigator
Masking Description: At the screening visit, all subjects will be randomly assigned a unique subject number (e.g., 001,002,003, etc.). Enrolled subjects will retain the subject number assigned at Screening Visit throughout the study. In phase Ib, no randomization will be performed. All subjects will receive the therapy chosen by the treating physician.
  Patients enrolled in phase II will be randomized through the application built in the eCRF in RedCap® for this purpose. Participant, care provider and Investigator will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metastatic gastrointestinal tumors and acute leukemia patients (Experimental): Patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and bile ducts) and newly diagnosed/relapse acute leukemias who meet the inclusion criteria will take the anamu extract with chemotherapy to evaluate the adverse drug-related side effects.
  Interventions: Drug: Petiveria Alliacea Preparation
- Stage II Metastatic gastrointestinal tumors including pancreas (Experimental): For solid metastatic tumors, 30 patients will be recruited, which can be from the colon, pancreas, stomach, and bile ducts, divided into two groups of 15 patients, an intervention group and a placebo group. The intervention group will receive the Esperanza extract at DMT for three continuous treatment cycles (approximately 12 weeks), and the other group will receive the placebo.
  Interventions: Drug: Petiveria Alliacea Preparation
- Stage II Placebo Metastatic gastrointestinal tumors including pancreas (Placebo Comparator): For solid metastatic tumors, 30 patients will be recruited, which can be from the colon, pancreas, stomach, and bile ducts, divided into two groups of 15 patients, an intervention group and a placebo group. The intervention group will receive the Esperanza extract at DMT for three continuous treatment cycles (approximately 12 weeks), and the other group will receive the placebo. Both groups will receive standard chemotherapy treatment for their underlying disease. The safety evaluation will be carried out in each treatment cycle, and the efficacy evaluation will be carried out at the end of the three cycles.
  Interventions: Drug: Placebo
- Acute leukemia (Newly/Relapse) (Experimental): For newly diagnosed hematological tumors, 28 patients will be recruited and will receive the Esperanza extract at DMT. The intervention group will continuously receive the Esperanza extract at DMT for four weeks with the standard chemotherapy regimen for their underlying disease. The safety and efficacy evaluation will be carried out at the end of the treatment cycle.
  Patients with relapsed or refractory acute leukemias will be admitted to receive the calculated DMT in phase Ib; A total of 6 patients will be recruited, and safety and efficacy evaluations will be performed during three treatment cycles or progression and death of the patient.
  For the analysis of the response in patients with acute leukemia, a comparison will be made with a group followed historically. A propensity score matching will be performed for statistical analysis in case of differences in their baseline characteristics.
  Interventions: Drug: Petiveria Alliacea Preparation

INTERVENTIONS:
Drug: Petiveria Alliacea Preparation — Petiveria Alliacea Preparation in pill
  Arms: Acute leukemia (Newly/Relapse); Metastatic gastrointestinal tumors and acute leukemia patients; Stage II Metastatic gastrointestinal tumors including pancreas
Drug: Placebo — Placebo in pill
  Arms: Stage II Placebo Metastatic gastrointestinal tumors including pancreas

SUMMARY:
This is a phase Ib/II clinical study that has two phases. In phase Ib, the safety evaluation of the extract of Petiveria alliacea (Esperanza) will be carried out in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and biliary tract) and patients with newly diagnosed and relapsed acute leukemia. In phase IIb, the safety will continue to be evaluated, and the efficacy of the Esperanza extract will be explored in combination with chemotherapy in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and biliary tract) with newly diagnosed acute leukemias and relapses.

DETAILED DESCRIPTION:
Anamú, Petiveria alliacea, has been used by traditional medicine to treat leukemia and breast cancer. However, its activity on tumor metabolism makes it a therapeutic candidate for many tumors with alterations in glycolytic metabolism, but also uses the mitochondria to produce energy.

Given the glycolytic nature of some tumor cells, the modulating activity of cell metabolism exerted by anamú extract may be partly responsible for the anti-tumor activity.

Previous reports show that some patients with ALL or AML whose response to treatment was evaluated in vitro are sensitive to a standardized extract of Petiveria alliacea. Even more interesting is the fact that when we treat the cells with allopathic therapy, explicitly established for each of these pathologies, the sensitivity of the blasts increases when they are treated concomitantly with the extract, which suggests that the intrinsic resistance of each one of tumor cells in the different tissues evaluated can be reduced by the action of the phytomedicine. The same thing was observed when spheres obtained from human breast cancer were co-treated with the anamú extract and anthracyclines. These observations allow to validate the traditional use of anamú in the treatment of some tumors, such as leukemia and breast cancer, among others. However, to observe the safety and effects on patients, it is necessary to develop a clinical study that would allow the anamú phytomedicine produced in the appropriate pharmaceutical conditions, to be included as a complementary therapy based on a standardized extract of the plant and that can overcome the resistance of tumor cells to conventional treatments, improving response and increasing overall survival of patients in Colombia.

Although the explosion of new therapies in solid tumors and hematological alterations is not so high, countries such as Germany, France, and Italy have used traditional medicine from which herbal pharmaceutical preparations are derived in the treatment of different types of diseases, including cancer. , estimating the use of these products between 30 and 75% of patients worldwide. These herbal products are mainly used to reduce allopathic therapies' side effects and organic toxicity, protect and stimulate the immune system, or prevent future neoplasms or their recurrence. Currently, various extracts from natural products are in clinical trials in the United States, and there is significant evidence about some plants' role in leukemia's evolution.

This is a phase Ib/II clinical study that has two phases. In phase Ib, the safety evaluation of the extract of Petiveria alliacea (Esperanza) will be carried out in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and biliary tract) and patients with newly diagnosed and relapsed acute leukemia. In phase IIb, the safety will continue to be evaluated, and the efficacy of the Esperanza extract will be explored in combination with chemotherapy in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and biliary tract) with newly diagnosed acute leukemias and relapses.

ELIGIBILITY:
Inclusion Criteria Solid Tumors:

1. Patients must be over 18 years of age, with no upper age limit
2. Histological diagnosis of gastrointestinal cancer may include stomach, colon, bile ducts, and pancreas.
3. Measurable disease through diagnostic tests and who will receive chemotherapy as primary treatment for their disease.
4. At least one discrete metastatic site identified
5. ECOG scale status from 0 to 2 with survival more significant than two months.
6. Subject can swallow and retain oral medication and does not have uncontrolled emesis or persistent diarrhea.
7. Adequate renal, hematological, hepatic, and cardiac function at the investigator's discretion.
8. Without uncontrolled or significant comorbidities determined by clinical history, physical examination, and screening laboratories at the investigator's discretion.
9. Patients of childbearing age and without safe non-hormonal planning methods must have a negative pregnancy test before the screening.
10. Fertile female subjects (those who have not been postmenopausal for at least 12 months or are surgically sterile by bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and their male partners must use at least one of the contraceptive methods listed below during study entry, throughout the study, and for at least six months after use of the P2Et extract (the effects of the P2Et extract on the developing human fetus are unknown):

a. Complete abstinence from sexual intercourse, beginning at least one complete menstrual cycle before administration of study drug; (It should be noted: sexual abstinence as a contraceptive method should be limited to those cases where it is already established as the patient's pre-existing lifestyle choice).

b. Vasectomy in the partner of a female subject c. Intrauterine device (IUD) d. Double-barrier method (condom, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jelly or cream).

k) Desire to complete the study and follow-up interventions.

Inclusion Criteria Acute Leukemia:

1. Patients must be over 18 years of age, with no upper age limit
2. Patients who have had a new diagnosis of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) will be eligible for the study and are eligible for chemotherapy treatment.

   * Patients must be newly diagnosed
   * Patients must have failed initial therapy, which may manifest in any of the following ways:

     * Demonstration of primary refractory disease (primary induction failure) as evidenced by mid-cycle bone marrow analysis showing lack of complete tumor clearance (CTC).
     * Relapse of the initial disease after a period of achieving complete remission.
3. Subject can swallow and retain oral medication and does not have uncontrolled emesis or persistent diarrhea.
4. Adequate renal, hematological, and hepatic function at the investigator's discretion.
5. Without uncontrolled or significant comorbidities determined by clinical history, physical examination, and screening laboratories at the investigator's discretion.
6. Patients of childbearing age and without safe non-hormonal planning, methods must have a negative pregnancy test before the screening.
7. Fertile female subjects (those who have not been postmenopausal for at least 12 months or are surgically sterile by bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and their male partners must use at least one of the contraceptive methods listed below. Listed below during study entry, throughout the study, and for at least six months after use of the P2Et extract (the effects of the P2Et extract on the developing human fetus are unknown):

a. Complete abstinence from sexual intercourse, beginning at least one complete menstrual cycle before administration of study drug; (It should be noted: sexual abstinence as a contraceptive method should be limited to those cases where it is already established as the patient's pre-existing lifestyle choice).

b. Vasectomy in the partner of a female subject c. Intrauterine device (IUD) d. Double-barrier method (condom, contraceptive sponge, diaphragm, or vaginal ring with spermicidal jelly or cream).

h) Desire to complete the study and follow-up interventions.

Exclusion Criteria:

The exclusion criteria apply to solid tumors as well as hematological tumors.

Subjects with one or more conditions are not eligible for this study.

1. Subjects treated in any other therapeutic clinical protocol 30 days prior to study entry or during study participation.
2. Patients receiving other investigational agents.
3. The female subject is pregnant or nursing. A negative serum or urine pregnancy test obtained at screening should confirm that the woman is not pregnant. Pregnancy tests are not required for postmenopausal or surgically sterilized women.
4. Serious concomitant morbidity, active at the discretion of the investigator
5. Subjects with a confirmed diagnosis of HIV before enrollment or a positive diagnosis of HIV at the time of screening.
6. Recipients of solid organ transplants.
7. Any condition that, in the opinion of the principal investigator, makes the subject ineligible to participate in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy | 12 months
  Evaluate the adverse drug reactions of cancer patients treated with anamú extract and chemotherapy through the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Quality of life in patients | 12 months
  Changes of at least 5 points above the difference between the groups of the functional scales of the patients evaluated using the EORTC QLQ-C-30 scale
Tumor response | 12 months
  To determine the impact of treatment with Esperanza extract in combination with chemotherapy on the number and size of metastases.
Survival | 12 months
  To determine event/progression-free survival in patients with metastatic gastrointestinal tumors (colon, pancreas, stomach, and bile ducts) and patients with newly diagnosed and relapsed acute leukemias.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Di Martino MT, Zazzeroni F, Donadelli M, Chiodoni C, Caraglia M, Scotlandi K, Meschini S, Leonetti C. Reprogramming Tumor-Immune Cell Interface in Solid and Hematological Malignancies to Enhance Response to Therapy. J Exp Clin Cancer Res. 2018 Mar 5;37(1):48. doi: 10.1186/s13046-018-0710-x. No abstract available. PMID 29506548
- [Result] Uruena C, Sandoval TA, Lasso P, Tawil M, Barreto A, Torregrosa L, Fiorentino S. Evaluation of chemotherapy and P2Et extract combination in ex-vivo derived tumor mammospheres from breast cancer patients. Sci Rep. 2020 Nov 12;10(1):19639. doi: 10.1038/s41598-020-76619-9. PMID 33184339
- [Result] Sharma SV, Lee DY, Li B, Quinlan MP, Takahashi F, Maheswaran S, McDermott U, Azizian N, Zou L, Fischbach MA, Wong KK, Brandstetter K, Wittner B, Ramaswamy S, Classon M, Settleman J. A chromatin-mediated reversible drug-tolerant state in cancer cell subpopulations. Cell. 2010 Apr 2;141(1):69-80. doi: 10.1016/j.cell.2010.02.027. PMID 20371346
- [Result] Bergers G, Fendt SM. The metabolism of cancer cells during metastasis. Nat Rev Cancer. 2021 Mar;21(3):162-180. doi: 10.1038/s41568-020-00320-2. Epub 2021 Jan 18. PMID 33462499
- [Result] Fong MY, Zhou W, Liu L, Alontaga AY, Chandra M, Ashby J, Chow A, O'Connor ST, Li S, Chin AR, Somlo G, Palomares M, Li Z, Tremblay JR, Tsuyada A, Sun G, Reid MA, Wu X, Swiderski P, Ren X, Shi Y, Kong M, Zhong W, Chen Y, Wang SE. Breast-cancer-secreted miR-122 reprograms glucose metabolism in premetastatic niche to promote metastasis. Nat Cell Biol. 2015 Feb;17(2):183-94. doi: 10.1038/ncb3094. Epub 2015 Jan 26. PMID 25621950
- [Result] Eddy RJ, Weidmann MD, Sharma VP, Condeelis JS. Tumor Cell Invadopodia: Invasive Protrusions that Orchestrate Metastasis. Trends Cell Biol. 2017 Aug;27(8):595-607. doi: 10.1016/j.tcb.2017.03.003. Epub 2017 Apr 12. PMID 28412099
- [Result] Kang X, Wang J, Li C. Exposing the Underlying Relationship of Cancer Metastasis to Metabolism and Epithelial-Mesenchymal Transitions. iScience. 2019 Nov 22;21:754-772. doi: 10.1016/j.isci.2019.10.060. Epub 2019 Oct 31. PMID 31739095
- [Result] Xian ZY, Liu JM, Chen QK, Chen HZ, Ye CJ, Xue J, Yang HQ, Li JL, Liu XF, Kuang SJ. Inhibition of LDHA suppresses tumor progression in prostate cancer. Tumour Biol. 2015 Sep;36(10):8093-100. doi: 10.1007/s13277-015-3540-x. Epub 2015 May 16. PMID 25983002
- [Result] Zhu J, Ma J, Wang X, Ma T, Zhang S, Wang W, Zhou X, Shi J. High Expression of PHGDH Predicts Poor Prognosis in Non-Small Cell Lung Cancer. Transl Oncol. 2016 Dec;9(6):592-599. doi: 10.1016/j.tranon.2016.08.003. PMID 27916294
- [Result] Butler LM, Perone Y, Dehairs J, Lupien LE, de Laat V, Talebi A, Loda M, Kinlaw WB, Swinnen JV. Lipids and cancer: Emerging roles in pathogenesis, diagnosis and therapeutic intervention. Adv Drug Deliv Rev. 2020;159:245-293. doi: 10.1016/j.addr.2020.07.013. Epub 2020 Jul 23. PMID 32711004
- [Result] Shah US, Dhir R, Gollin SM, Chandran UR, Lewis D, Acquafondata M, Pflug BR. Fatty acid synthase gene overexpression and copy number gain in prostate adenocarcinoma. Hum Pathol. 2006 Apr;37(4):401-9. doi: 10.1016/j.humpath.2005.11.022. Epub 2006 Feb 7. PMID 16564913
- [Result] Koundouros N, Poulogiannis G. Reprogramming of fatty acid metabolism in cancer. Br J Cancer. 2020 Jan;122(1):4-22. doi: 10.1038/s41416-019-0650-z. Epub 2019 Dec 10. PMID 31819192
- [Result] Itkonen HM, Brown M, Urbanucci A, Tredwell G, Ho Lau C, Barfeld S, Hart C, Guldvik IJ, Takhar M, Heemers HV, Erho N, Bloch K, Davicioni E, Derua R, Waelkens E, Mohler JL, Clarke N, Swinnen JV, Keun HC, Rekvig OP, Mills IG. Lipid degradation promotes prostate cancer cell survival. Oncotarget. 2017 Jun 13;8(24):38264-38275. doi: 10.18632/oncotarget.16123. PMID 28415728
- [Result] Zadra G, Photopoulos C, Tyekucheva S, Heidari P, Weng QP, Fedele G, Liu H, Scaglia N, Priolo C, Sicinska E, Mahmood U, Signoretti S, Birnberg N, Loda M. A novel direct activator of AMPK inhibits prostate cancer growth by blocking lipogenesis. EMBO Mol Med. 2014 Apr;6(4):519-38. doi: 10.1002/emmm.201302734. Epub 2014 Feb 4. PMID 24497570
- [Result] Song K, Li M, Xu X, Xuan LI, Huang G, Liu Q. Resistance to chemotherapy is associated with altered glucose metabolism in acute myeloid leukemia. Oncol Lett. 2016 Jul;12(1):334-342. doi: 10.3892/ol.2016.4600. Epub 2016 May 17. PMID 27347147
- [Result] Song K, Li M, Xu XJ, Xuan L, Huang GN, Song XL, Liu QF. HIF-1alpha and GLUT1 gene expression is associated with chemoresistance of acute myeloid leukemia. Asian Pac J Cancer Prev. 2014;15(4):1823-9. doi: 10.7314/apjcp.2014.15.4.1823. PMID 24641416
- [Result] Herst PM, Howman RA, Neeson PJ, Berridge MV, Ritchie DS. The level of glycolytic metabolism in acute myeloid leukemia blasts at diagnosis is prognostic for clinical outcome. J Leukoc Biol. 2011 Jan;89(1):51-5. doi: 10.1189/jlb.0710417. Epub 2010 Oct 19. PMID 20959411
- [Result] Guerra F, Arbini AA, Moro L. Mitochondria and cancer chemoresistance. Biochim Biophys Acta Bioenerg. 2017 Aug;1858(8):686-699. doi: 10.1016/j.bbabio.2017.01.012. Epub 2017 Feb 1. PMID 28161329
- [Result] Bokil A, Sancho P. Mitochondrial determinants of chemoresistance. Cancer Drug Resist. 2019 Sep 19;2(3):634-646. doi: 10.20517/cdr.2019.46. eCollection 2019. PMID 35582564
- [Result] Panina SB, Baran N, Brasil da Costa FH, Konopleva M, Kirienko NV. A mechanism for increased sensitivity of acute myeloid leukemia to mitotoxic drugs. Cell Death Dis. 2019 Aug 13;10(8):617. doi: 10.1038/s41419-019-1851-3. PMID 31409768
- [Result] Sriskanthadevan S, Jeyaraju DV, Chung TE, Prabha S, Xu W, Skrtic M, Jhas B, Hurren R, Gronda M, Wang X, Jitkova Y, Sukhai MA, Lin FH, Maclean N, Laister R, Goard CA, Mullen PJ, Xie S, Penn LZ, Rogers IM, Dick JE, Minden MD, Schimmer AD. AML cells have low spare reserve capacity in their respiratory chain that renders them susceptible to oxidative metabolic stress. Blood. 2015 Mar 26;125(13):2120-30. doi: 10.1182/blood-2014-08-594408. Epub 2015 Jan 28. PMID 25631767
- [Result] Yang J, Ren B, Yang G, Wang H, Chen G, You L, Zhang T, Zhao Y. The enhancement of glycolysis regulates pancreatic cancer metastasis. Cell Mol Life Sci. 2020 Jan;77(2):305-321. doi: 10.1007/s00018-019-03278-z. Epub 2019 Aug 20. PMID 31432232
- [Result] Donadelli M, Dando I, Dalla Pozza E, Palmieri M. Mitochondrial uncoupling protein 2 and pancreatic cancer: a new potential target therapy. World J Gastroenterol. 2015 Mar 21;21(11):3232-8. doi: 10.3748/wjg.v21.i11.3232. PMID 25805929
- [Result] Lu W, Hu Y, Chen G, Chen Z, Zhang H, Wang F, Feng L, Pelicano H, Wang H, Keating MJ, Liu J, McKeehan W, Wang H, Luo Y, Huang P. Novel role of NOX in supporting aerobic glycolysis in cancer cells with mitochondrial dysfunction and as a potential target for cancer therapy. PLoS Biol. 2012;10(5):e1001326. doi: 10.1371/journal.pbio.1001326. Epub 2012 May 8. PMID 22589701
- [Derived] Ballesteros-Ramirez R, Pinilla P, Sanchez J, Arevalo M, Sanchez E, Aschner P, Uruena C, Fiorentino S. Exploring the safety and efficacy of phytomedicine Petiveria alliacea extract (Esperanza) in patients with metastatic gastrointestinal tumors and acute leukemias: study protocol for a phase Ib/randomized double blind phase II trial (PA001). BMC Complement Med Ther. 2023 Aug 10;23(1):284. doi: 10.1186/s12906-023-04109-2. PMID 37563608